CLINICAL TRIAL: NCT01167829
Title: Pharmacokinetics of Modified Slow-Release Oral Testosterone Over 10 Days in Normal Men With Experimental Hypogonadism
Brief Title: ORAL T-8 Oral Testosterone for Male Hormonal Contraception
Acronym: Oral T8
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, John Amory, Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 38636-D
Record Dates: First submitted 2010-07-20; First posted 2010-07-22 (Estimated); Results first posted 2013-08-23 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-08

CONDITIONS: Healthy
Keywords: Experimental; Acyline plus 27 oral testosterone pills; taken 3x/day
MeSH Terms: interventions — Testosterone; acyline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acyline and oral testosterone (Experimental)
  Interventions: Drug: Oral Testosterone; Drug: Acyline

INTERVENTIONS:
Drug: Oral Testosterone — Oral Testosterone: 300 mg, pills, three times daily Day 1 - 10 (total of 27 pills)
Drug: Acyline — 300 ug/kg injection on Day 0

SUMMARY:
The purpose of this study is to test how the body absorbs a new form of oral testosterone (T). On Day 1 and Day 9 there are overnight stays in the General Clinical Research Center at the University of Washington to monitor blood testosterone levels over a 24-hour period.

DETAILED DESCRIPTION:
We will administer two experimental drugs, acyline and oral testosterone. Acyline shots will be given on Day 0 to turn off the body's testosterone production for about 10-14 days.

The next day, Day 1, subjects begin taking 300 mg modified slow-release testosterone pill by mouth, three times a day, around 9 AM, 1 PM, and 7 PM for a total of 27 pills.

There are overnight stays on Day 1 and Day 9 to allow monitoring of blood testosterone levels over a 24 hour period, from @9 AM to 9 AM the next morning. At those visits, blood is drawn at baseline (before taking the pill) and at 1, 2, 4, 5, 6, 8, 10, 11, 12, 14, 16, and 24 hours after the morning dose.

Acyline is an experimental drug. The FDA allows its use only in research with a small number of volunteers. We have used acyline in over 125 men without serious side effects. The use of testosterone in this study is experimental and there may be unknown or unanticipated risks.

ELIGIBILITY:
INCLUSION CRITERIA:

* able and willing to
* not participate in another drug study or donate blood, not take medications
* use contraception, comply with the protocol

EXCLUSION CRITERIA:

* abnormal evaluation, based on physical exam, medical history, blood tests (including serum chemistry, hematology, HIV, HCV, hormone levels)
* history or current use of alcohol, drug, steroid abuse, >3 alcohol drinks/day
* history of testicular disease, severe testicular trauma, major psychiatric disorder, bleeding disorders, current use of anti-coagulants or testosterone
* participation in hormonal drug study within past month

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2010-07; Primary Completion 2010-10 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John K Amory, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Background] Katznelson L, Finkelstein JS, Schoenfeld DA, Rosenthal DI, Anderson EJ, Klibanski A. Increase in bone density and lean body mass during testosterone administration in men with acquired hypogonadism. J Clin Endocrinol Metab. 1996 Dec;81(12):4358-65. doi: 10.1210/jcem.81.12.8954042.
- [Background] Behre HM, Kliesch S, Leifke E, Link TM, Nieschlag E. Long-term effect of testosterone therapy on bone mineral density in hypogonadal men. J Clin Endocrinol Metab. 1997 Aug;82(8):2386-90. doi: 10.1210/jcem.82.8.4163. PMID 9253305
- [Background] Bhasin S, Bremner WJ. Clinical review 85: Emerging issues in androgen replacement therapy. J Clin Endocrinol Metab. 1997 Jan;82(1):3-8. doi: 10.1210/jcem.82.1.3640. No abstract available. PMID 8989221
- [Background] Wang C, Alexander G, Berman N, Salehian B, Davidson T, McDonald V, Steiner B, Hull L, Callegari C, Swerdloff RS. Testosterone replacement therapy improves mood in hypogonadal men--a clinical research center study. J Clin Endocrinol Metab. 1996 Oct;81(10):3578-83. doi: 10.1210/jcem.81.10.8855804.
- [Background] Snyder PJ, Peachey H, Berlin JA, Hannoush P, Haddad G, Dlewati A, Santanna J, Loh L, Lenrow DA, Holmes JH, Kapoor SC, Atkinson LE, Strom BL. Effects of testosterone replacement in hypogonadal men. J Clin Endocrinol Metab. 2000 Aug;85(8):2670-7. doi: 10.1210/jcem.85.8.6731. PMID 10946864
- [Background] Kelch RP, Jenner MR, Weinstein R, Kaplan SL, Grumbach MM. Estradiol and testosterone secretion by human, simian, and canine testes, in males with hypogonadism and in male pseudohermaphrodites with the feminizing testes syndrome. J Clin Invest. 1972 Apr;51(4):824-30. doi: 10.1172/JCI106877. PMID 4259253
- [Background] Weinstein RL, Kelch RP, Jenner MR, Kaplan SL, Grumbach MM. Secretion of unconjugated androgens and estrogens by the normal and abnormal human testis before and after human chorionic gonadotropin. J Clin Invest. 1974 Jan;53(1):1-6. doi: 10.1172/JCI107526. PMID 4271572
- [Background] Herbst KL, Anawalt BD, Amory JK, Bremner WJ. Acyline: the first study in humans of a potent, new gonadotropin-releasing hormone antagonist. J Clin Endocrinol Metab. 2002 Jul;87(7):3215-20. doi: 10.1210/jcem.87.7.8675. PMID 12107227
- [Background] Herbst KL, Coviello AD, Page S, Amory JK, Anawalt BD, Bremner WJ. A single dose of the potent gonadotropin-releasing hormone antagonist acyline suppresses gonadotropins and testosterone for 2 weeks in healthy young men. J Clin Endocrinol Metab. 2004 Dec;89(12):5959-65. doi: 10.1210/jc.2003-032123. PMID 15579744
- [Background] Bagatell CJ, Bremner WJ. Androgens in men--uses and abuses. N Engl J Med. 1996 Mar 14;334(11):707-14. doi: 10.1056/NEJM199603143341107. No abstract available. PMID 8594431
- [Background] Fossa SD, Opjordsmoen S, Haug E. Androgen replacement and quality of life in patients treated for bilateral testicular cancer. Eur J Cancer. 1999 Aug;35(8):1220-5. doi: 10.1016/s0959-8049(99)00123-9. PMID 10615233
- [Background] Swerdloff RS, Wang C, Cunningham G, Dobs A, Iranmanesh A, Matsumoto AM, Snyder PJ, Weber T, Longstreth J, Berman N. Long-term pharmacokinetics of transdermal testosterone gel in hypogonadal men. J Clin Endocrinol Metab. 2000 Dec;85(12):4500-10. doi: 10.1210/jcem.85.12.7045. PMID 11134099
- [Background] Snyder CN, Clark RV, Caricofe RB, Bush MA, Roth MY, Page ST, Bremner WJ, Amory JK. Pharmacokinetics of 2 novel formulations of modified-release oral testosterone alone and with finasteride in normal men with experimental hypogonadism. J Androl. 2010 Nov-Dec;31(6):527-35. doi: 10.2164/jandrol.109.009746. Epub 2010 Apr 8. PMID 20378927
- [Background] de Ronde W. Hyperandrogenism after transfer of topical testosterone gel: case report and review of published and unpublished studies. Hum Reprod. 2009 Feb;24(2):425-8. doi: 10.1093/humrep/den372. Epub 2008 Oct 23. PMID 18948313
- [Background] Brachet C, Vermeulen J, Heinrichs C. Children's virilization and the use of a testosterone gel by their fathers. Eur J Pediatr. 2005 Oct;164(10):646-7. doi: 10.1007/s00431-005-1714-z. Epub 2005 Jul 16. PMID 16025298
- [Background] Amory JK, Matsumoto AM. The therapeutic potential of testosterone patches. Expert Opin Investig Drugs. 1998 Dec;7(12):1977-85. doi: 10.1517/13543784.7.12.1977. PMID 15991940
- [Background] 1. Plymate SR "Male Hypogonadism" in Principles and Practice of Endocrinology and Metabolism (3rd. Ed). Ed. Kenneth Becker, pp:1125-1150

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited through news media (website)and college campus bulletin boards in Seattle, WA. between July-September 2010. All visits were at the University of Washington, Seattle, WA.
Pre-assignment Details: 14 subjects were screened and 2 did not meet inclusion criteria for untreated high blood pressure and peripheral arterial disease.
Groups:
- Acyline and 0ral Testosterone: Acyline 300 mcg/kg subcutaneous + 300mg modified slow-release oral testosterone tid
Period: Overall Study
Arm/Group | Acyline and 0ral Testosterone
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Acyline and Oral Testosterone: 300 mcg/kg acyline, and modified slow-release oral testosterone 300 mg
Arm/Group | Acyline and Oral Testosterone
Number analyzed (Participants) | 12
Age Continuous [Median (Inter-Quartile Range); unit: years] | 28.1 [19 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 12
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.2 (1.5)
Body Weight [Mean (Standard Deviation); unit: kg] | 79.9 (7.5)
Follicle-stimulating hormone (FSH) [Mean (Standard Deviation); unit: IU/L] | 3.2 (1.5)
Luteinizing hormone (LH) [Mean (Standard Deviation); unit: IU/L] | 5.4 (4.4)
Testosterone [Mean (Standard Deviation); unit: ng/dL] | 510 (13)
Prostate-specific antigen (PSA) [Mean (Standard Deviation); unit: ng/mL] | 0.91 (0.56)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Testosterone Concentration
Description: initial pharmacokinetics [PK] (day 1) of oral testosterone dosed 3 times daily and the PK after 9 days of treatment
Time Frame: baseline & day 9
Population: per protocol
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/dL
Groups:
- Acyline and 300 mg Oral Testosterone: 300 mg oral testosterone three times daily
Arm/Group | Acyline and 300 mg Oral Testosterone
Number analyzed (Participants) | 12
ng/dL
  Day 1 | 924 (44)
  Day 9 | 741 (71)
Statistical Analysis 1: Comparison: Acyline and 300 mg Oral Testosterone; Test type: Superiority or Other; p = 0.05, t-test, 2 sided; Mean Difference (Net) = 183, Standard Error of Mean 44

2. Primary Outcome: Mean Testosterone Concentration
Description: initial 24-hour pharmacokinetics (PK) of oral testosterone dosed 3 times daily and post 24-hour PK after 9 days of treatment
Time Frame: baseline & day 9
Population: per protocol
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/dL
Groups:
- Acyine and 300 mg Oral Testosterone: 300 mg oral testosterone three times daily
Arm/Group | Acyine and 300 mg Oral Testosterone
Number analyzed (Participants) | 12
ng/dL
  Day 1 | 378 (45)
  Day 9 | 315 (41)

3. Secondary Outcome: Maximum Dihydrotestosterone (DHT) Concentration
Time Frame: baseline & day 9
Population: per protocol
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/dL
Groups:
- 300 mg Oral Testosterone: 300 mg oral testosterone three times daily
Arm/Group | 300 mg Oral Testosterone
Number analyzed (Participants) | 12
ng/dL
  Day 1 | 233 (49)
  Day 9 | 142 (55)

4. Secondary Outcome: Mean Dihydrotestosterone (DHT) Concentration
Time Frame: baseline & day 9
Population: per protocol
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/dL
Arm/Group | Acyline and 300 mg Oral Testosterone
Number analyzed (Participants) | 12
ng/dL
  Day 1 | 96 (38)
  Day 9 | 69 (41)

5. Secondary Outcome: Maximum Sex Hormone-Binding Globulin (SHGB)Concentration
Time Frame: baseline & day 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/dL
Arm/Group | 300 mg Oral Testosterone
Number analyzed (Participants) | 12
ng/dL
  Day 1 | 31 (48)
  Day 9 | 22 (48)

6. Secondary Outcome: Mean SHGB Concentration
Time Frame: baseline & day 9
Population: per protocol
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/dL
Arm/Group | 300 mg Oral Testosterone
Number analyzed (Participants) | 12
ng/dL
  Day 1 | 27 (46)
  Day 9 | 19 (14)

7. Secondary Outcome: Maximum Estradiol Concentration
Time Frame: baseline & day 9
Population: per protocol
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/dL
Arm/Group | 300 mg Oral Testosterone
Number analyzed (Participants) | 12
ng/dL
  Day 1 | 14 (28)
  Day 9 | 9 (27)

8. Secondary Outcome: Mean Estradiol Concentration
Time Frame: baseline & day 9
Population: per protocol
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/dL
Arm/Group | 300 mg Oral Testosterone
Number analyzed (Participants) | 12
ng/dL
  Day 1 | 11 (18)
  Day 9 | 7 (18)

9. Secondary Outcome: Free T Maximum Concentration
Description: Free T normal range 4.7-18 ng/dL
Time Frame: baseline & day 9
Population: per protocol
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/dL
Arm/Group | 300 mg Oral Testosterone
Number analyzed (Participants) | 12
ng/dL
  Day 1-2 | 24 (47)
  Day 9-10 | 21 (86)

10. Secondary Outcome: Free Testosterone Mean Concentration
Description: Free T normal range 4.7-18 ng/dL
Time Frame: baseline & day 9
Population: per protocol
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/dL
Arm/Group | 300 mg Oral Testosterone
Number analyzed (Participants) | 12
ng/dL
  Day 1-2 | 8.7 (43)
  Day 9-10 | 8.3 (37)

ADVERSE EVENTS:
Time Frame: 4 months, July - October 2010
Description: The first subject was screened 7/13/2010; the last subject exited 10/25/2010. Subjects in the study are asked about adverse events and concomitant medications at every visit.
Arm/Group | Acyline and Oral Testosterone
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 8/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acyline and Oral Testosterone (N=12)
hypogonadal symptoms (Endocrine disorders) | 1 (1) — low libido, irritability
Headache (General disorders) | 1 (1)
upper respiratory infection (Infections and infestations) | 2 (2)
confusion (General disorders) | 1 (1) — transient episode likely due to heat exposure
musculoskeletal injury (Musculoskeletal and connective tissue disorders) | 2 (2)
elevated serum aspartate aminotrasferase (Investigations) | 1 (1) — day 4 of treatment
elevated serum alanine aminotransferase (Investigations) | 1 (1) — day 4 of treatment
elevated serum bilirubin (Investigations) | 1 (1) — day 4 of treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes